CLINICAL TRIAL: NCT05858398
Title: Influence of Body Composition, Total Body Fat and Body Mass Index on the Pharmacokinetics of Docetaxel in Localized Breast Cancer
Brief Title: Influence of Body Composition on Chemotherapy Outcomes in Localized Breast Cancer
Acronym: FATTAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Collaborators: Erasmus Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB22.03
Record Dates: First submitted 2023-04-14; First posted 2023-05-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; body composition; docetaxel; pharmacokinetics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmocokinetics blood sample assessment (Experimental): during first administration of docetaxel several pharmacokinetics samples will be assessed
  Interventions: Biological: pharmacokinetics blood sample assessment

INTERVENTIONS:
Biological: pharmacokinetics blood sample assessment — pharmacokinetics blood sample assessment during the first exposure to docetaxel

SUMMARY:
The purpose of this study is to determine if pharmacokinetics of docetaxel is modified by the body composition (assessed by the BMI but also by CT-scan) in patients treated by docetaxel as adjuvant treatment of a localized breast cancer

DETAILED DESCRIPTION:
Half of the patients treated for a localized breast cancer are obese or overweighted. Recently published post-hoc analyses of a large randomised trial (BIG-2-98) revealed that BMI could impact the benefit of a docetaxel based chemotherapy, but not of an anthracyclin based chemotherapy.

One of the hypothesis is that the distribution volume of hydrophobic drugs, such as docetaxel, may be influenced by the BMI, and more precisely by the amount of total fat.

In that context, we aim to assess the docetaxel pharmacokinetics during its first exposure for localized breast cancer, and compare these results according to 3 groups of patients (lean, overweight and obese).

ELIGIBILITY:
Inclusion Criteria:

* Woman older than
* Early breast cancer
* CT-scan of less than 3 months, including L3 level
* Indication of docetaxel at 100 mg/m² as adjuvant CT

Exclusion Criteria:

* HER2 amplified or triple negative tumors
* Pregnant or breastfeeding women
* Patients under guardianship or curatorship
* Concomitant administration of another cytotoxic drug or targeted therapy
* Psychosocial disorder
* Administration of another cytotoxic drug or targeted therapy within 20 days prior to blood collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of docetaxel area under courb between obese and lean patients | 8 hours after the end of first cycle of docetaxel

SECONDARY OUTCOMES:
Comparison of docetaxel area under courb between overweight and lean patients | 8 hours after the end of first cycle of docetaxel
Comparison of docetaxel area under courb according to BMI versus body composition (assessed by CT scan) | 8 hours after the end of first cycle of docetaxel
Interrelationship of docetaxel area under courb and docetaxel induced side effects | 3 months after first cycle of docetaxel
Interrelationship between of body composition and leptine/adiponectine rates | 8 hours after the end of first cycle of docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Florian Clatot, Prof, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No